CLINICAL TRIAL: NCT04547361
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of E2511 in Healthy Subjects
Brief Title: A Study to Assess the Safety and Tolerability of E2511 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: E2511-A001-004
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteers
Keywords: E2511; Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1: Dose 1 E2511 or Placebo (Experimental): Participants will receive Dose 1 of E2511 or E2511 matched placebo, tablets, orally, once on Day 1 under fasted condition.
  Interventions: Drug: E2511; Drug: E2511 Matched Placebo
- Cohort 2: Dose 2 E2511 or Placebo (Experimental): Participants will receive Dose 2 of E2511 or E2511 matched placebo, tablets, orally, once on Day 1 under fasted condition.
  Interventions: Drug: E2511; Drug: E2511 Matched Placebo
- Cohort 3: Dose 3 E2511 or Placebo (Experimental): Participants will receive Dose 3 of E2511 or E2511 matched placebo, tablets, orally, once on Day 1 (Treatment Period 1) under fasted condition followed by Dose 3 of E2511 or E2511 matched placebo, tablets, orally, once on Day 7 (Treatment Period 2) under fed condition. A washout period of 6 days will be maintained between the doses.
  Interventions: Drug: E2511; Drug: E2511 Matched Placebo
- Cohort 4: Dose 4 E2511 or Placebo (Experimental): Participants will receive Dose 4 of E2511 or E2511 matched placebo, tablets, orally, once on Day 1 under fasted condition.
  Interventions: Drug: E2511; Drug: E2511 Matched Placebo
- Cohort 5: Dose 5 E2511 or Placebo (Experimental): Participants will receive Dose 5 of E2511 or E2511 matched placebo, tablets, orally, once on Day 1 under fasted condition.
  Interventions: Drug: E2511; Drug: E2511 Matched Placebo
- Cohort 6: Dose 6 E2511 or Placebo (Experimental): Participants will receive Dose 6 of E2511 or E2511 matched placebo, tablets, orally, once on Day 1 under fasted condition.
  Interventions: Drug: E2511; Drug: E2511 Matched Placebo
- Cohort 7: Dose 3 E2511 (Elderly Participants) or Placebo (Experimental): Elderly participants will receive Dose 3 of E2511 or E2511 matched placebo, tablets, orally, once on Day 1 under fasted condition.
  Interventions: Drug: E2511; Drug: E2511 Matched Placebo

INTERVENTIONS:
Drug: E2511 — E2511 tablets.
Drug: E2511 Matched Placebo — Placebo tablets matching E2511 tablets.

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability, and pharmacokinetic (PK) of E2511 following single ascending oral doses in healthy adult and elderly participants.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking, age greater than or equal to (>=) 18 years and less than (<) 55 years old adult male or female (Cohorts 1 - 6) or age >=65 years and less than or equal to (<=) 85 years old elderly male or female (Cohort 7) at the time of informed consent
2. Weight of at least 50 kilogram (kg) and body mass index >=18 and <30 kilogram per square meter (kg/m^2) at Screening

Exclusion Criteria:

1. Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria (that is, not of childbearing potential or practicing highly effective contraception throughout the study period plus 90 days after study drug discontinuation). No sperm donation is allowed during the study period plus 90 days after discharge from the study.
2. Females who are breastfeeding or pregnant at Screening or Baseline
3. Females of childbearing potential who:

   * Within 28 days before study entry, did not use a highly effective method of contraception,
   * Do not agree to use a highly effective method of contraception (as described above) throughout the entire study period and for 28 days after study drug discontinuation.
4. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
5. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing
6. Evidence of disease related to chronic headaches, migraines, joint pain or other disorders or disease resulting in chronic or intermittent pain within 4 weeks before dosing
7. Any personal or family history of seizures (including febrile seizures) or diagnosis of epilepsy or episode of unexplained loss of consciousness
8. Any history of neurological or other medical conditions which in the opinion of the investigator has the potential to reduce seizure threshold
9. Any epileptiform discharges in EEG at Screening
10. A prolonged QT/ QT interval corrected for heart rate (QTc) interval >450 millisecond [ms]) A history of risk factors for torsade de pointes
11. History of prolonged QT/QTc interval
12. Left bundle branch block
13. History of myocardial infarction or active ischemic heart disease
14. History of clinically significant arrhythmia or uncontrolled arrhythmia
15. Any lifetime history of suicidal ideation or any lifetime history of suicidal behavior as indicated by the C-SSRS
16. Any lifetime history of psychiatric disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Cohorts 1, 2, 3, 4, 5, 6, 7: Number of Participants Reporting one or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From screening up to 28 days after last dose of study drug (up to 63 days)
Cohorts 1, 2, 3, 4, 5, 6, 7: Number of Participants With Markedly Abnormal Laboratory Values | From screening up to 28 days after last dose of study drug (up to 63 days)
Cohorts 1, 2, 3, 4, 5, 6, 7: Number of Participants With Clinically Significant Change From Screening in Vital Signs Values | From screening up to 28 days after last dose of study drug (up to 63 days)
Cohorts 1, 2, 3, 4, 5, 6, 7: Number of Participants With Clinically Significant Change From Screening in Electrocardiograms (ECGs) Findings | From screening up to 28 days after last dose of study drug (up to 63 days)
Cohorts 1, 2, 3, 4, 5, 6, 7: Number of Participants With Treatment-emergent Suicidal Ideation or Suicidal Behavior as Measured Using Columbia-Suicide Severity Rating Scale (C-SSRS) | From screening up to 28 days after last dose of study drug (up to 63 days)
  The C-SSRS (mapped to Columbia Classification Algorithm of Suicide Assessment [C-CASA]) is an interview-based rating scale to systematically assess any suicidality, suicidal behavior, or suicidal ideation. Any suicidality is emergence of any suicidal ideation or suicidal behavior. Any suicidal behavior is indicated when response is "yes" for any these questions- actual attempt to suicide, engaged in non-suicidal self-injurious behavior, interrupted attempt, aborted attempt, preparatory acts. Any suicidal ideation is indicated when response is "yes" for any of these questions- wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent to suicide.
Cohorts 1, 2, 3, 4, 5, 6, 7: Number of Participants With Clinically Significant Change From Screening in Physical Examination Findings | From screening up to 28 days after last dose of study drug (up to 63 days)
Cohorts 1, 2, 3, 4, 5, 6, 7: Number of Participants With Clinically Significant Change From Screening in Neurological Exam Findings | Cohorts 1, 2, 4, 5, 6, 7: Screening up to Day 1 (approximately 28 days); Cohort 3: Screening up to Day 7 (approximately 35 days)
Cohorts 1, 2, 3, 4, 5, 6, 7: Number of Participants With Clinically Significant Change From Screening in Psychiatric Assessment | From screening up to 28 days after last dose of study drug (up to 63 days)
  Number of participants with clinically significant change in psychiatric assessment will be evaluated by a psychiatrist as a measure of mental health assessment.
Cohorts 1, 2, 3, 4, 5, 6, 7: Number of Participants With Clinically Significant Change From Screening in Electroencephalogram (EEG) Measurements | From screening up to Day 2 (approximately 30 days)
Cohorts 1, 2, 3, 4, 5, 6, 7: Maximum Observed Plasma Concentration (Cmax) for E2511 on Day 1 | Day 1: pre-dose up to a potential maximum of 120 hours post-dose
Cohort 3: Maximum Observed Plasma Concentration (Cmax) for E2511 on Day 7 | Day 7: pre-dose up to a potential maximum of 120 hours post-dose
Cohorts 1, 2, 3, 4, 5, 6, 7: Time to Reach Cmax (tmax) for E2511 on Day 1 | Day 1: pre-dose up to a potential maximum of 120 hours post-dose
Cohort 3: Time to Reach Cmax (tmax) for E2511 on Day 7 | Day 7: pre-dose up to a potential maximum of 120 hours post-dose
Cohorts 1, 2, 3, 4, 5, 6, 7: Area Under the Plasma Concentration-time Curve (AUC(0-t)) From Time Zero to the Last Quantifiable Plasma Concentration for E2511 on Day 1 | Day 1: pre-dose up to a potential maximum of 120 hours post-dose
Cohort 3: Area Under the Plasma Concentration-time Curve (AUC(0-t)) From Time Zero to the Last Quantifiable Plasma Concentration for E2511 on Day 7 | Day 7: pre-dose up to a potential maximum of 120 hours post-dose
Cohorts 1, 2, 3, 4, 5, 6, 7: Area Under the Plasma Concentration-time Curve (AUC(0-inf)) From Time Zero to Infinity for E2511 on Day 1 | Day 1: pre-dose up to a potential maximum of 120 hours post-dose
Cohort 3: Area Under the Plasma Concentration-time Curve (AUC(0-inf)) From Time Zero to Infinity for E2511 on Day 7 | Day 7: pre-dose up to a potential maximum of 120 hours post-dose
Cohorts 1, 2, 3, 4, 5, 6, 7: Area Under the Plasma Concentration-time Curve (AUC(0-24)) From Time Zero to 24 Hours Postdose for E2511 on Day 1 | Day 1: pre-dose up to a potential maximum of 24 hours post-dose
Cohort 3: Area Under the Plasma Concentration-time Curve (AUC(0-24)) From Time Zero to 24 Hours Postdose for E2511 on Day 7 | Day 7: pre-dose up to a potential maximum of 24 hours post-dose
Cohorts 1, 2, 3, 4, 5, 6, 7: Terminal Elimination Phase Half-Life (t1/2) for E2511 on Day 1 | Day 1: pre-dose up to a potential maximum of 120 hours post-dose
Cohort 3: Terminal Elimination Phase Half-Life (t1/2) for E2511 on Day 7 | Day 7: pre-dose up to a potential maximum of 120 hours post-dose
Cohorts 1, 2, 3, 4, 5, 6, 7: Apparent Total Clearance (CL/F) for E2511 on Day 1 | Day 1: pre-dose up to a potential maximum of 120 hours post-dose
Cohort 3: Apparent Total Clearance (CL/F) for E2511 on Day 7 | Day 7: pre-dose up to a potential maximum of 120 hours post-dose
Cohorts 1, 2, 3, 4, 5, 6, 7: Apparent Volume of Distribution at Terminal Phase (Vz/F) for E2511 on Day 1 | Day 1: pre-dose up to a potential maximum of 120 hours post-dose
Cohort 3: Apparent Volume of Distribution at Terminal Phase (Vz/F) for E2511 on Day 7 | Day 7: pre-dose up to a potential maximum of 120 hours post-dose

SECONDARY OUTCOMES:
Cohort 3: Geometric Mean Ratio of Cmax Between the Fasted and Fed State for E2511 20 mg | Days 1 and 7: pre-dose up to a potential maximum of 120 hours post-dose
Cohort 3: Geometric Mean Ratio of AUC(0-t) Between the Fasted and fed State for E2511 20 mg | Days 1 and 7: pre-dose up to a potential maximum of 120 hours post-dose
Cohort 3: Geometric Mean Ratio of AUC(0-inf) Between the Fasted and fed State for E2511 20 mg | Days 1 and 7: pre-dose up to a potential maximum of 120 hours post-dose
Cohort 3 and Cohort 7: Geometric Mean Ratio of Cmax Between the Healthy Elderly and Adult Participants for E2511 20 mg | Cohort 3: Days 1 and 7: pre-dose up to a potential maximum of 120 hours post-dose; Cohort 7: Day 1: pre-dose up to a potential maximum of 120 hours post-dose
Cohort 3 and Cohort 7: Geometric Mean Ratio of AUC(0-t) Between the Healthy Elderly and Adult Participants for E2511 20 mg | Cohort 3: Days 1 and 7: pre-dose up to a potential maximum of 120 hours post-dose; Cohort 7: Day 1: pre-dose up to a potential maximum of 120 hours post-dose
Cohort 3 and Cohort 7: Geometric Mean Ratio of AUC(0-inf) Between the Healthy Elderly and Adult Participants for E2511 20 mg | Cohort 3: Days 1 and 7: pre-dose up to a potential maximum of 120 hours post-dose; Cohort 7: Day 1: pre-dose up to a potential maximum of 120 hours post-dose
Cohorts 1, 2, 3, 4, 5, 6, 7: Correlation Between QTc and E2511 Plasma Concentrations | Day 1: Pre-dose through 24 hours post dose
  To explore the correlation between changes in QTc interval (msec) and E2511 plasma concentrations, appropriate correction method for QTc interval calculation such as QTcF will used for analysis. Holter monitors will be used to collect continuous 12-lead ECG data, from which high precision ECG recordings will be extracted from the Holter monitor data prior to the PK blood samples collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.